CLINICAL TRIAL: NCT05184543
Title: Effects of Different Exercise Programs on Injury Risk and Sports Performance in Adolescent Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ETK00-2021-0086
Record Dates: First submitted 2022-01-05; First posted 2022-01-11 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Sport Injury
Keywords: Injury prevention; Exercise; Sports performance; Basketball; Warm up
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Participants in the control group will continue their routine warm-up programs.
  Interventions: Other: Routine Exercise Program
- Core Stability Group (Experimental): A warm-up program including core stability exercises will be applied to the participants.
  Interventions: Other: Core Stability Exercise Program
- Neuromuscular Exercise Group (Experimental): A warm-up program including dynamic neuromuscular exercises will be applied to the participants.
  Interventions: Other: Body Weight Neuromuscular Warm-Up Program

INTERVENTIONS:
Other: Routine Exercise Program — 8 weeks of routine basketball training will be done. Dynamic stretching exercises, in which large muscle groups are exercised, can be applied for 20 minutes.
  Arms: Control Group
Other: Core Stability Exercise Program — In addition to the 8-week routine basketball training, 20 min core stability exercises will be given to the Core Group. Core stability exercises will be performed on the stable surface for the first 4 weeks, and core stability exercises will be performed on unstable surfaces for the next 4 weeks.
  Arms: Core Stability Group
Other: Body Weight Neuromuscular Warm-Up Program — Each 20-minute program consists of 5 different parts. The beginning of the program consists of low-speed running exercises with the ball. The running track for each exercise will include 4 basketball court areas. The second part consists of active stretching exercises. The third part consists of exercises focusing on general strength. The fourth part consists of plyometric, balance, and jump exercises. The final section consists of a sprint with sudden changes of direction and basketball movements.
  Arms: Neuromuscular Exercise Group

SUMMARY:
Basketball is a team sport where aerobic and anaerobic performance is important. Knowing how to reduce common injuries and risk is important when designing a warm-up exercise program for basketball. Various warm-up programs, including neuromuscular training, are thought to reduce the incidence of lower extremity injuries and improve athletic performance in athletes. There are several neuromuscular training programs designed to improve joint position sense, increase joint stability, develop protective joint reflexes, and ultimately prevent lower extremity injuries. In the literature, there is a need for studies comparing the effects of various warm-up programs applied to adolescent licensed basketball players on injury risks and basketball-specific sportive performance parameters. Therefore, the aim of the study is to examine the effects of different exercise programs on injury risk and sportive performance in adolescent basketball players.

DETAILED DESCRIPTION:
Basketball is a team sport where aerobic and anaerobic performance is important. Knowing how to reduce common injuries and risk is important when designing a basketball training program. It has been stated that injuries in basketball are injuries caused by muscle imbalances.

Various warm-up programs, including neuromuscular training, have been shown to reduce the incidence of lower extremity injuries in athletes. Various neuromuscular training programs designed to improve joint position sense, increase joint stability, develop protective joint reflexes, and ultimately prevent lower extremity injuries have been explored.

According to Zazulak et al, a lack of neuromuscular control of body core muscles can lead to uncontrolled trunk displacement during movement. Core strength is very important for many sports, including basketball, athletics, football, and jumping, to maintain correct posture and to perform some daily activities such as walking, climbing stairs, and stepping. Strong core stability helps in transferring high muscle strength. Core muscle function can affect structures from the waist to the ankle, and deficiencies in core muscle capacity can increase the risk of lower extremity injury.

In a study by Sannicandro et al in 2020, in which they examined the effect of core stability exercises added to the warm-up program in prepubertal basketball players on sprint and jump performances, they showed that there was an improvement in jump and sprint performances as a result of training given for 4 weeks and 2 sessions per week.

Benis et al. In 2017, in a study examining the effects of neuromuscular training with bodyweight on Y-balance test (YBT) performances in elite female basketball players; It was observed that there was an improvement in YBT scores after the 8-week program. The program included a sport-specific neuromuscular warm-up designed to improve athletic performance and prevent lower extremity injuries. Based on these findings, a neuromuscular training program called the "Italian Basketball Injury Prevention Program" was developed.

Bonato, Benis et al. In the study where they examined the effects of a neuromuscular training program, which included lower extremity strength, agility, jumping, and general exercises with the ball, which were included in the routine warm-up program in 2017, on the prevention of lower extremity injuries in elite female basketball players during the regular season; It has been stated that the incidence of lower extremity injuries has decreased.

Functional movement definition is also very important for athletes. Functional movement is the ability to generate and maintain a balance between mobility and stability along the kinetic chain while performing basic movement patterns with accuracy and efficiency. Performance-based mobility-competence-based tests have been established in recent years to identify deficits in neuromuscular status associated with increased risk of injury. In this context, it has been seen that the most commonly used tests in the literature are Functional Movement Screen (FMS), Y balance test (YBT), trunk stabilization tests, and jump tests.

When investigators look at the literature, there is a need to investigate various warm-up programs that reduce the risk of injury in adolescent licensed basketball players and investigate their effects on explosive strength, speed, agility, and balance parameters, which are essential for basketball. In this study, in addition to the routine warm-up program consisting of programs in which muscle groups are dynamically stretched, one group only included core stabilization exercises; The other group will be given programs that include exercises to be done with the ball and neuromuscular warm-up exercises with body weight.

ELIGIBILITY:
Inclusion Criteria:

* To be a female licensed basketball player between the ages of 12-18.
* To train regularly and as a team at least 3 days a week.

Exclusion Criteria:

* History of any lower extremity injury and surgery in the 6 months prior to the study.
* Not participating in regular and team training at least 3 days a week during the working process.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen | 10 weeks
  Functional Movement Analysis (FMS) will be used to determine the risk of injury and functional movement. Identification of movement disorders assists clinicians in the preparation and implementation of an appropriate rehabilitation program following injuries and the development of injury prevention plans. FMS consists of 7 subtests including the deep squat, high stepping, cross stepping, shoulder mobility, active straight leg raise, trunk stability, rotational stability. It is stated that there is a risk of injury below 14 points, with a maximum of 21 points.

SECONDARY OUTCOMES:
Vertical Jump | 10 weeks
  The vertical jump height of the athletes will be measured by Microgate optojump® (Microgate, Bolzano, Italy) device. The OptoJump device is a device that has been studied for reliability. Athletes' jumps from the ground up were recorded in cm. The greater the amount of bounce, the better the test. Vertical jump tests will be performed as 1 exercise and then 2 tests, and the test result with a better score than 2 correct measurements will be used in statistical analysis. In this test, hands-free active jumping will be performed.
Horizontal Jump | 10 weeks
  A horizontal jump test will be used the upper body and arms are rotated to assist in jumping, and both legs are brought closer together before starting the jump. After the jump, the descent is made on both sides and the distance from the heel to the starting point is measured. Distances are standardized as distance/height according to the height of the participants. 2 attempts were taken and the best score was recorded.
Sprint | 10 weeks
  The 30 m sprint test will be used to evaluate the speed. 30 m determined points are adjusted with photocells. The participant exits the determined point at full speed and the test is completed when the photocell is passed after 30 m. The time is recorded in seconds (17). Microgate Witty wireless training timer will be used as the device.
Agility | 10 weeks
  Agility will be evaluated with the T-test. A test platform is established with 4 cones. There is a distance of 10m between the two cones in the middle and between the two cones placed on the sides. The participant quickly runs 10 meters around the cone and goes to the cone on the left. He turns from there and runs to the next right cone. Then the test is completed when it comes to the middle cone again and runs to the starting point. Measurements are made with the help of photocells at the starting point. The time is recorded in seconds. It will be done with the Microgate Witty wireless training timer device.
Lower Quarter Balance | 10 weeks
  The balance will be evaluated with the Y balance test for the lower extremity. Participants' leg lengths will be measured from the anterior supra iliac to the distal of the medial malleolus. First, the participants will be required to try reaching out in each direction 6 times. They will be asked to lie down 3 times in each direction and will be recorded in centimeters. If the weight is transferred to the reaching foot, if the fixed foot is separated from the floor and the hands are separated from the hips, it will be considered an error and the test will be repeated. Scores calculated with "Best Reach / Leg Length) x 100 = % max reach" for each direction will be normalized. The total score will be calculated by averaging the normalized anterolateral, posterolateral, and posteromedial scores.

CONTACTS AND LOCATIONS:
Overall Officials: Tayfun ARSLAN, Specialist Physiotherapist, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Atatürk Spor Salonu, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No